CLINICAL TRIAL: NCT03601013
Title: Demographical and Clinical Profile of Patients on Dual Antıplatelet Therapy and Mean Precise-DAPT and DAPT Scores in Turkey
Status: Completed | Type: Observational
Sponsor: Cardiovascular Academy Society, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: DAPT-TR
Record Dates: First submitted 2018-03-27; First posted 2018-07-26 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Anti-platelet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Demographical and Clinical Profile of Patients on Dual Antıplatelet Therapy — Demographical and Clinical Profile of Patients on Dual Antıplatelet Therapy

SUMMARY:
Coronary Artery Disease (CAD) is leading cause of death worldwide. Most of them underwent coronary angiography and they have to use dual anti-platelet therapy. As mentioned novel guidelines for CAD, the estimated number of patients requiring dual anti-platelet therapy has increased over time, and DAPT time is controversial. Acting on the behalf of 2017 ESC focused update on dual anti-platelet therapy in coronary artery disease developed in collaboration with EACTS guideline, this study is amid to determine PRECISE-DAPT score which predicts out of hospital bleeding risk in patients receiving dual anti-platelet treatment and to detect the prevalence of patients with high bleeding risk, and to determine DAPT score which predicts benefit/risk ratio of continuing or discontinuing dual ant-iplatelet therapy after 12 months and to detect the prevalence of patients with high ischemic or hemorrhagic complication risk in centers included in this study.

DETAILED DESCRIPTION:
Design

The study is a national, multicenter, non-interventional, observational, prospective registry.

Population

Patients older than 18 years old of age, have acute coronary syndrome or percutaneous coronary intervention electively and with available admission hemoglobin, white blood cell and creatine clearance data will be enrolled for Precise-DAPT,and Patients older than 18 years old of age and completed 12 months of dual anti-platelet therapy without having hemorrhage and ischemic coronary event and with available data of age, history of smoking, presence of diabetes mellitus, history of percutaneous coronary intervention, paclitaxel eluting stent, stent diameter, history of myocardial infarction, saphenous vein graft intervention, ejection fraction or presence of heart failure. Patients that do not approve informed consent will be excluded.

Aim

This study is amid to investigate the demographic and clinical profile of patients with CAD and on dual anti-platelet therapy, mean precise -DAPT and DAPT scores of Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have acute coronary syndrome or percutaneous coronary intervention electively and with available admission heamoglobin, white blood cell and creatine clearance data and on dual antiplatelet therapy

Exclusion Criteria:

* Being under eighteen years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have acute coronary syndrome or percutaneous coronary intervention electively and with available admission heamoglobin, white blood cell and creatine clearance data and on dual antiplatelet therapy
Sampling Method: Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
ischemia | 3 months
  ischemic events of patients on dual antiplatelet therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No